CLINICAL TRIAL: NCT02210923
Title: Carotid Baroreflex Activation and Its Effect on the Chemoreflex Study
Brief Title: Effect Baroreflex Activation Therapy on the Carotid Body
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: CVRx, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NL3770006813
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Hypertension Resistant To Conventional Therapy; Baroreflex; Carotid Body
Keywords: Baroreflex; Electrical stimulation; Carotid body; Chemoreceptors; Resistant hypertension
MeSH Terms: conditions — Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood for analysis of PaCO2, PaO2 and pH
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Resistant hypertensive patients with Rheos system: We will program 6 electrical device activation setting twice in a random order to see what happens with the aforementioned respiratory and cardiovascular variables. The following electrical settings will be programmed for 4 minutes each setting:
  * 20 Hz, 3 Volts, 480 microseconds
  * 20 Hz, 6 Volts, 480 microseconds
  * 50 Hz, 3 Volts, 480 microseconds
  * 50 Hz, 6 Volts, 480 microseconds
  * 90 Hz, 3 Volts, 480 microseconds
  * 90 Hz, 6 Volts, 480 microseconds

SUMMARY:
Carotid baroreflex activation therapy (BAT) by the Rheos® system produces a sustained fall in blood pressure in patients with resistant hypertension. Since the activation electrodes are implanted at the level of the carotid sinus, it is conceivable that the nearby located carotid body chemoreceptors are stimulated as well. Physiological stimulation of carotid chemoreceptors not only raises respiration, but it also increases sympathetic activity which may in part counteract the effects of BAT. The aim of the present study is to investigate whether there is evidence for concomitant carotid chemoreflex activation during BAT. We hypothesized that there is no clinically relevant co-activation of the carotid body chemoreceptors during BAT in patients with resistant hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Be currently implanted with Rheos system and have completed the 13-month follow-up period.
* Be on stable anti-hypertensive therapy for at least 4 weeks prior to inclusion, where stable is defined as no changes in medications or dosage of medications.
* Have at least one functional carotid baroreflex activation electrode.
* Have signed and approved informed consent form for participation in this study.

Exclusion Criteria:

* Myocardial infarction (MI) or cerebral vascular accident (CVA) within the past 90 days, or subject is still unstable from a prior MI or CVA that occurred more than 90 days ago.
* Are unable or unwilling to comply with the protocol requirements of this study.
* Diagnosed with severe chronic obstructive lung disease (COPD/asthma GOLD stadium III and IV).

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects implanted with a BAT system will be invited to participate in this study. These are patients who were enrolled in the DEBuT-HET and Rheos Pivotal Trial and have given their permission to be approached for follow-up studies. Subjects are all >21 years of age and were all known with a blood pressure ≥160/90 mmHg despite optimal antihypertensive therapy before receiving BAT. It is essential to have the Rheos® device implanted to enable participation in this study, as we want to investigate the effect of electrical carotid sinus activation on the carotid body chemoreflex.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in arterial CO2 (PaCO2) during baroreflex activation therapy | 6 times during different electrical activation settings within one hour
  During one hour several device activation settings will be programmed at random. During each device setting we will collect arterial blood samples to check for PaCO2.

SECONDARY OUTCOMES:
Change in end-tidal CO2 during baroreflex activation therapy | 1 - 1.25 hour
  Change in respiratory variables will be analyzed during the aforementioned time frame in which we will program several device activation settings.
Change in blood pressure during baroreflex activation therapy | 1 - 1.25 hour
  The change in cardiovascular variables will be analyzed during each device activation setting
Change in respiratory rate during baroreflex activation therapy | 1 - 1.25 hour
  Change in respiratory variables will be analyzed during the aforementioned time frame in which we will program several device activation settings.
Change in expiration time during baroreflex activation therapy | 1 - 1.25 hour
  Change in respiratory variables will be analyzed during the aforementioned time frame in which we will program several device activation settings.
Change in heart rate during baroreflex activation therapy | 1 - 1.25 hour
  The change in cardiovascular variables will be analyzed during each device activation setting
Change in peripheral vascular resistance during baroreflex activation therapy | 1 - 1.25 hour
  The change in cardiovascular variables will be analyzed during each device activation setting
Change in forced expiratory volume-1 second (FEV1) before and after turning off the device | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Abraham Kroon, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center+, Maastricht, Netherlands

REFERENCES:
- See also: Overall description of the device and related safety and efficacy results — http://cvrx.com